CLINICAL TRIAL: NCT04331145
Title: REACTIC-TAVI Trial: Platelet REACtivity According to TICagrelor Dose After Transcatheter AorticValve Implantation. A Pilot Study.
Brief Title: Platelet REACtivity According to TICagrelor Dose After Transcatheter AorticValve Implantation
Acronym: REACTIC-TAVI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andres Iñiguez Romo (Other)
Responsible Party: Sponsor-Investigator, Andres Iñiguez Romo, MD, phD, Fundacin Biomedica Galicia Sur
Organization: Fundacin Biomedica Galicia Sur (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REACTIC2019-HAC; 2019-004860-23 (EudraCT Number)
Record Dates: First submitted 2020-03-24; First posted 2020-04-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Symptomatic Aortic Stenosis
Keywords: Transcatheter aortic valve implantation (TAVI); Transcatheter aortic valve replacement (TAVR); Antiplatelet therapy; Ticagrelor; Clopidogrel
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clopidogrel 75 mg (No Intervention): Platelet reactivity will be assessed by VerifyNow P2Y12 assay in ALL enrolled patients after confirmed use of clopidogrel for 4 days prior TAVI. Patients that have not completed a pre-treatment period of 4 days of clopidogrel will receive a loading dose of 300mg, according to the clinical practice, with assessment of platelet reactivity by VerifyNow P2Y12 at the following 6 hours. Based on results of basal VerifyNow P2Y12 assay at least 24 hours before the index-TAVI procedure, patients with:
  Normal basal platelet reactivity (PRU < 160 assessed with VerifyNow P2Y12 assay): Patients will continue with clopidogrel 75 mg/day until TAVI and during the following three months. All patients will be assessed by clinical follow up and platelet reactivity according to the protocol. Prescription of aspirin 100mg/day will be encourage as per guidelines recommendations.
- Ticagrelor 60 mg (Active Comparator): Platelet reactivity will be assessed by VerifyNow P2Y12 assay in ALL enrolled patients after confirmed use of clopidogrel for 4 days prior TAVI. Patients that have not completed a pre-treatment period of 4 days of clopidogrel will receive a loading dose of 300mg, according to the clinical practice, with assessment of platelet reactivity by VerifyNow P2Y12 at the following 6 hours. Based on results of basal VerifyNow P2Y12 assay at least 24 hrs before the index-TAVI procedure, patients with:
  High on-treatment platelet reactivity (PRU ≥ 160 assessed with VerifyNow P2Y12 assay): Patients will be switched to receive ticagrelor 60mg twice daily initiating at least 24 hours before TAVI procedure, in order to arrive to the index TAVI procedure with at least two doses of 60 mg, and will continue with Ticagrelor 60mg twice per day during the following three months.
  Interventions: Drug: Ticagrelor 60mg

INTERVENTIONS:
Drug: Ticagrelor 60mg — Platelet reactivity will be assessed by VerifyNow P2Y12 assay in ALL enrolled patients after confirmed use of clopidogrel for 4 days prior TAVI. Patients that have not completed a pre-treatment period of 4 days of clopidogrel will receive a loading dose of 300mg, according to the clinical practice, with assessment of platelet reactivity by VerifyNow P2Y12 at the following 6 hours. Based on results of basal VerifyNow P2Y12 assay at least 24 hours before the index-TAVI procedure, patients with:
  High on-treatment platelet reactivity (PRU ≥ 160 assessed with VerifyNow P2Y12 assay): Patients will be switched to receive ticagrelor 60mg twice daily initiating at least 24hrs before TAVI procedure, in order to arrive to the index TAVI procedure with at least two doses of 60 mg, and will continue with Ticagrelor 60mg twice per day during the following three months.
  Other Names: High platelet reactivity patients
  Arms: Ticagrelor 60 mg

SUMMARY:
The narrowing of the aortic valve, which prevents blood from reaching the entire body correctly is a common disease in our environment. To correct this problem, many patients undergo Transcatheter Aortic Valve Implantation (TAVI) according to standard clinical practice. Patients have to continue with a specific pharmacological treatment (antiplatelet agents) to avoid possible complications during the first months after the procedure. This treatment is not yet well established. Current guidelines recommend dual antiplatelet therapy with Aspirin and Clopidogrel for 3-6 months after TAVI to avoid thromboembolic complications. But the risk of bleeding events with DAPT in this population is not negligible.

This study aims to determine the degree of response to Ticagrelor 60 mg every 12 hours as a single antiplatelet strategy in patients who do not achieve an adequate response with Clopidogrel 75mg every 24 hours. The study will evaluate if patients have an adequate response to Clopidogrel and if not, then patients will start treatment with Ticagrelor 60 mg every 12 hours after TAVI and until completing 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe symptomatic aortic stenosis
* Accepted for transfemoral TAVI by a Heart Team decision
* Evaluation of platelet reactivity assessed by VerifyNow® assay prior TAVI

Exclusion Criteria:

* Contraindication to TAVI
* TAVI performed by a different access route than transfemoral
* Ned for oral anticoagulation therapy
* History of intracranial hemorrhage
* Ischemic stroke the 14 days before TAVI
* Active pathological bleeding or diathesis
* Moderate to severe hepatic impairment
* Use of strong CYP34A inhibitors or inducers
* Contraindications to DAPT for 3 months
* Contraindication to clopidogrel or ticagrelor
* Platelet count <50,000
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment in suppressing High Platelet Reactivity | At least 24 hours before the index-TAVI procedure
  Assess the efficacy of ticagrelor 60 mg/12 hours in suppressing High Platelet Reactivity after TAVI. Platelet reactivity will be assessed by VerifyNow P2Y12.
Efficacy of treatment in suppressing High Platelet Reactivity | 24 ± 2 hour post TAVI
  Assess the efficacy of ticagrelor 60 mg/12 hours in suppressing High Platelet Reactivity after TAVI. Platelet reactivity will be assessed by VerifyNow P2Y12.
Efficacy of treatment in suppressing High Platelet Reactivity | 30 ± 7 days post TAVI
  Assess the efficacy of ticagrelor 60 mg/12 hours in suppressing High Platelet Reactivity after TAVI. Platelet reactivity will be assessed by VerifyNow P2Y12.
Efficacy of treatment in suppressing High Platelet Reactivity | 90 ± 7 days post TAVI
  Assess the efficacy of ticagrelor 60 mg/12 hours in suppressing High Platelet Reactivity after TAVI. Platelet reactivity will be assessed by VerifyNow P2Y12.

SECONDARY OUTCOMES:
Security: incidence of hemorrhagic complications | 1) At least 24 hours before the index-TAVI procedure 2) 3) 4) 5)
  Evaluate the incidence of hemorrhagic complications after TAVI. As safety endpoint we will assess the incidence of investigator-reported clinical events according to VARC-2 criteria (death, myocardial infarction, stroke, TIA, acute renal injury, bleeding, vascular access-site and access-related complications), including BARC bleeding definitions. For safety endpoint, all BARC criteria, included in VARC-2 criteria will be recorded.
Security: incidence of hemorrhagic complications | 24 ± 2 hour post TAVI
  Evaluate the incidence of hemorrhagic complications after TAVI. As safety endpoint we will assess the incidence of investigator-reported clinical events according to VARC-2 criteria (death, myocardial infarction, stroke, TIA, acute renal injury, bleeding, vascular access-site and access-related complications), including BARC bleeding definitions. For safety endpoint, all BARC criteria, included in VARC-2 criteria will be recorded.
Security: incidence of hemorrhagic complications | 30 ± 7 days post TAVI
  Evaluate the incidence of hemorrhagic complications after TAVI. As safety endpoint we will assess the incidence of investigator-reported clinical events according to VARC-2 criteria (death, myocardial infarction, stroke, TIA, acute renal injury, bleeding, vascular access-site and access-related complications), including BARC bleeding definitions. For safety endpoint, all BARC criteria, included in VARC-2 criteria will be recorded.
Security: incidence of hemorrhagic complications | 90 ± 7 days post TAVI
  Evaluate the incidence of hemorrhagic complications after TAVI. As safety endpoint we will assess the incidence of investigator-reported clinical events according to VARC-2 criteria (death, myocardial infarction, stroke, TIA, acute renal injury, bleeding, vascular access-site and access-related complications), including BARC bleeding definitions. For safety endpoint, all BARC criteria, included in VARC-2 criteria will be recorded.
Security: incidence of hemorrhagic complications | 120 ± 7 days post TAVI
  Evaluate the incidence of hemorrhagic complications after TAVI. As safety endpoint we will assess the incidence of investigator-reported clinical events according to VARC-2 criteria (death, myocardial infarction, stroke, TIA, acute renal injury, bleeding, vascular access-site and access-related complications), including BARC bleeding definitions. For safety endpoint, all BARC criteria, included in VARC-2 criteria will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Victor A Jimenez Diaz, MD, MPH, Principal Investigator — Hospital Álvaro Cunqueiro
Locations (1):
- Hospital Alvaro Cunqueiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cannon CP, Husted S, Harrington RA, Scirica BM, Emanuelsson H, Peters G, Storey RF; DISPERSE-2 Investigators. Safety, tolerability, and initial efficacy of AZD6140, the first reversible oral adenosine diphosphate receptor antagonist, compared with clopidogrel, in patients with non-ST-segment elevation acute coronary syndrome: primary results of the DISPERSE-2 trial. J Am Coll Cardiol. 2007 Nov 6;50(19):1844-51. doi: 10.1016/j.jacc.2007.07.053. Epub 2007 Oct 23. PMID 17980250
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] James S, Akerblom A, Cannon CP, Emanuelsson H, Husted S, Katus H, Skene A, Steg PG, Storey RF, Harrington R, Becker R, Wallentin L. Comparison of ticagrelor, the first reversible oral P2Y(12) receptor antagonist, with clopidogrel in patients with acute coronary syndromes: Rationale, design, and baseline characteristics of the PLATelet inhibition and patient Outcomes (PLATO) trial. Am Heart J. 2009 Apr;157(4):599-605. doi: 10.1016/j.ahj.2009.01.003. PMID 19332184
- [Background] Toma N. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of Ticagrelor versus Clopidogrel in patients with stable coronary artery disease. The ONSET/OFFSET study. Maedica (Bucur). 2010 Jan;5(1):75-6. No abstract available. PMID 21977127
- [Background] Adams HP Jr. Ticagrelor, a new antiplatelet agent, for prevention of ischemic events in patients with coronary artery disease. Curr Neurol Neurosci Rep. 2010 Jan;10(1):4-6. doi: 10.1007/s11910-009-0082-x. No abstract available. PMID 20425218
- [Background] Steg PG, James S, Harrington RA, Ardissino D, Becker RC, Cannon CP, Emanuelsson H, Finkelstein A, Husted S, Katus H, Kilhamn J, Olofsson S, Storey RF, Weaver WD, Wallentin L; PLATO Study Group. Ticagrelor versus clopidogrel in patients with ST-elevation acute coronary syndromes intended for reperfusion with primary percutaneous coronary intervention: A Platelet Inhibition and Patient Outcomes (PLATO) trial subgroup analysis. Circulation. 2010 Nov 23;122(21):2131-41. doi: 10.1161/CIRCULATIONAHA.109.927582. Epub 2010 Nov 8. PMID 21060072
- [Background] Varenhorst C, Alstrom U, Scirica BM, Hogue CW, Asenblad N, Storey RF, Steg PG, Horrow J, Mahaffey KW, Becker RC, James S, Cannon CP, Brandrup-Wognsen G, Wallentin L, Held C. Factors contributing to the lower mortality with ticagrelor compared with clopidogrel in patients undergoing coronary artery bypass surgery. J Am Coll Cardiol. 2012 Oct 23;60(17):1623-30. doi: 10.1016/j.jacc.2012.07.021. Epub 2012 Sep 26. PMID 23021325
- [Background] Jeong YH, Bliden KP, Antonino MJ, Park KS, Tantry US, Gurbel PA. Usefulness of the VerifyNow P2Y12 assay to evaluate the antiplatelet effects of ticagrelor and clopidogrel therapies. Am Heart J. 2012 Jul;164(1):35-42. doi: 10.1016/j.ahj.2012.03.022. Epub 2012 Jun 13. PMID 22795280
- [Background] Theidel U, Asseburg C, Giannitsis E, Katus H. Cost-effectiveness of ticagrelor versus clopidogrel for the prevention of atherothrombotic events in adult patients with acute coronary syndrome in Germany. Clin Res Cardiol. 2013 Jun;102(6):447-58. doi: 10.1007/s00392-013-0552-7. Epub 2013 Mar 9. PMID 23474908
- [Background] Bergmeijer TO, Janssen PW, Schipper JC, Qaderdan K, Ishak M, Ruitenbeek RS, Asselbergs FW, van 't Hof AW, Dewilde WJ, Spano F, Herrman JP, Kelder JC, Postma MJ, de Boer A, Deneer VH, ten Berg JM. CYP2C19 genotype-guided antiplatelet therapy in ST-segment elevation myocardial infarction patients-Rationale and design of the Patient Outcome after primary PCI (POPular) Genetics study. Am Heart J. 2014 Jul;168(1):16-22.e1. doi: 10.1016/j.ahj.2014.03.006. Epub 2014 Mar 21. PMID 24952855
- [Background] Jeong KH, Cho JH, Woo JS, Kim JB, Kim WS, Lee TW, Kim KS, Ihm CG, Kim W. Platelet reactivity after receiving clopidogrel compared with ticagrelor in patients with kidney failure treated with hemodialysis: a randomized crossover study. Am J Kidney Dis. 2015 Jun;65(6):916-24. doi: 10.1053/j.ajkd.2014.11.023. Epub 2015 Jan 24. PMID 25622774
- [Background] Cho JR, Rollini F, Franchi F, DeGroat C, Bhatti M, Dunn EC, Ferrante E, Muniz-Lozano A, Suryadevara S, Zenni MM, Guzman LA, Bass TA, Angiolillo DJ. Pharmacodynamic Effects of Ticagrelor Dosing Regimens in Patients on Maintenance Ticagrelor Therapy: Results From a Prospective, Randomized, Double-Blind Investigation. JACC Cardiovasc Interv. 2015 Jul;8(8):1075-1083. doi: 10.1016/j.jcin.2015.02.022. Epub 2015 Jun 24. PMID 26117466
- [Background] Alexopoulos D, Perperis A, Koniari I, Karvounis H, Patsilinakos S, Ziakas A, Barampoutis N, Panagiotidis T, Akinosoglou K, Hahalis G, Xanthopoulou I. Ticagrelor versus high dose clopidogrel in ST-segment elevation myocardial infarction patients with high platelet reactivity post fibrinolysis. J Thromb Thrombolysis. 2015 Oct;40(3):261-7. doi: 10.1007/s11239-015-1183-9. PMID 25680893
- [Background] Thomas MR, Outteridge SN, Ajjan RA, Phoenix F, Sangha GK, Faulkner RE, Ecob R, Judge HM, Khan H, West LE, Dockrell DH, Sabroe I, Storey RF. Platelet P2Y12 Inhibitors Reduce Systemic Inflammation and Its Prothrombotic Effects in an Experimental Human Model. Arterioscler Thromb Vasc Biol. 2015 Dec;35(12):2562-70. doi: 10.1161/ATVBAHA.115.306528. Epub 2015 Oct 29. PMID 26515417
- [Background] Andell P, James SK, Cannon CP, Cyr DD, Himmelmann A, Husted S, Keltai M, Koul S, Santoso A, Steg PG, Storey RF, Wallentin L, Erlinge D; PLATO Investigators. Ticagrelor Versus Clopidogrel in Patients With Acute Coronary Syndromes and Chronic Obstructive Pulmonary Disease: An Analysis From the Platelet Inhibition and Patient Outcomes (PLATO) Trial. J Am Heart Assoc. 2015 Oct 9;4(10):e002490. doi: 10.1161/JAHA.115.002490. PMID 26452988
- [Background] Magnani G, Storey RF, Steg G, Bhatt DL, Cohen M, Kuder J, Im K, Aylward P, Ardissino D, Isaza D, Parkhomenko A, Goudev AR, Dellborg M, Kontny F, Corbalan R, Medina F, Jensen EC, Held P, Braunwald E, Sabatine MS, Bonaca MP. Efficacy and safety of ticagrelor for long-term secondary prevention of atherothrombotic events in relation to renal function: insights from the PEGASUS-TIMI 54 trial. Eur Heart J. 2016 Jan 21;37(4):400-8. doi: 10.1093/eurheartj/ehv482. Epub 2015 Oct 5. PMID 26443023
- [Background] Storey RF, Angiolillo DJ, Bonaca MP, Thomas MR, Judge HM, Rollini F, Franchi F, Ahsan AJ, Bhatt DL, Kuder JF, Steg PG, Cohen M, Muthusamy R, Braunwald E, Sabatine MS. Platelet Inhibition With Ticagrelor 60 mg Versus 90 mg Twice Daily in the PEGASUS-TIMI 54 Trial. J Am Coll Cardiol. 2016 Mar 15;67(10):1145-1154. doi: 10.1016/j.jacc.2015.12.062. PMID 26965534
- [Background] Velders MA, Abtan J, Angiolillo DJ, Ardissino D, Harrington RA, Hellkamp A, Himmelmann A, Husted S, Katus HA, Meier B, Schulte PJ, Storey RF, Wallentin L, Gabriel Steg P, James SK; PLATO Investigators. Safety and efficacy of ticagrelor and clopidogrel in primary percutaneous coronary intervention. Heart. 2016 Apr;102(8):617-25. doi: 10.1136/heartjnl-2015-308963. Epub 2016 Feb 4. PMID 26848185
- [Background] Windecker S, Tijssen J, Giustino G, Guimaraes AH, Mehran R, Valgimigli M, Vranckx P, Welsh RC, Baber U, van Es GA, Wildgoose P, Volkl AA, Zazula A, Thomitzek K, Hemmrich M, Dangas GD. Trial design: Rivaroxaban for the prevention of major cardiovascular events after transcatheter aortic valve replacement: Rationale and design of the GALILEO study. Am Heart J. 2017 Feb;184:81-87. doi: 10.1016/j.ahj.2016.10.017. Epub 2016 Oct 31. PMID 27892890
- [Background] Jilaihawi H, Asch FM, Manasse E, Ruiz CE, Jelnin V, Kashif M, Kawamori H, Maeno Y, Kazuno Y, Takahashi N, Olson R, Alkhatib J, Berman D, Friedman J, Gellada N, Chakravarty T, Makkar RR. Systematic CT Methodology for the Evaluation of Subclinical Leaflet Thrombosis. JACC Cardiovasc Imaging. 2017 Apr;10(4):461-470. doi: 10.1016/j.jcmg.2017.02.005. PMID 28385256
- [Background] Holm M, Tornvall P, Westerberg J, Rihan Hye S, van der Linden J. Ticagrelor pharmacokinetics and pharmacodynamics in patients with NSTEMI after a 180-mg loading dose. Platelets. 2017 Nov;28(7):706-711. doi: 10.1080/09537104.2016.1265921. Epub 2017 Feb 2. PMID 28150519
- [Background] Linke A, Chandrasekhar J, Sartori S, Lefevre T, van Belle E, Schaefer U, Tchetche D, Sardella G, Webb J, Colombo A, Windecker S, Vogel B, Farhan S, Sorrentino S, Sharma M, Snyder C, Asgar A, Dumonteil N, Tamburino C, Hink U, Violini R, Stella P, Bernstein D, Deliargyris E, Hengstenberg C, Baber U, Mehran R, Anthopoulos P, Dangas G; BRAVO-3 Investigators. Effect of valve design and anticoagulation strategy on 30-day clinical outcomes in transcatheter aortic valve replacement: Results from the BRAVO 3 randomized trial. Catheter Cardiovasc Interv. 2017 Nov 15;90(6):1016-1026. doi: 10.1002/ccd.27154. Epub 2017 Jul 19. PMID 28498562
- [Background] Collet JP, Berti S, Cequier A, Van Belle E, Lefevre T, Leprince P, Neumann FJ, Vicaut E, Montalescot G. Oral anti-Xa anticoagulation after trans-aortic valve implantation for aortic stenosis: The randomized ATLANTIS trial. Am Heart J. 2018 Jun;200:44-50. doi: 10.1016/j.ahj.2018.03.008. Epub 2018 Mar 10. PMID 29898848
- [Background] Van Mieghem NM, Unverdorben M, Valgimigli M, Mehran R, Boersma E, Baber U, Hengstenberg C, Shi M, Chen C, Saito S, Veltkamp R, Vranckx P, Dangas GD. Edoxaban Versus standard of care and their effects on clinical outcomes in patients having undergone Transcatheter Aortic Valve Implantation in Atrial Fibrillation-Rationale and design of the ENVISAGE-TAVI AF trial. Am Heart J. 2018 Nov;205:63-69. doi: 10.1016/j.ahj.2018.07.006. Epub 2018 Aug 29. PMID 30172099
- [Background] Mangieri A, Montalto C, Poletti E, Sticchi A, Crimi G, Giannini F, Latib A, Capodanno D, Colombo A. Thrombotic Versus Bleeding Risk After Transcatheter Aortic Valve Replacement: JACC Review Topic of the Week. J Am Coll Cardiol. 2019 Oct 22;74(16):2088-2101. doi: 10.1016/j.jacc.2019.08.1032. PMID 31623768
- [Result] Jimenez Diaz VA, Tello-Montoliu A, Moreno R, Cruz Gonzalez I, Baz Alonso JA, Romaguera R, Molina Navarro E, Juan Salvadores P, Paredes Galan E, De Miguel Castro A, Bastos Fernandez G, Ortiz Saez A, Fernandez Barbeira S, Raposeiras Roubin S, Ocampo Miguez J, Serra Penaranda A, Valdes Chavarri M, Cequier Fillat A, Calvo Iglesias F, Iniguez Romo A. Assessment of Platelet REACtivity After Transcatheter Aortic Valve Replacement: The REAC-TAVI Trial. JACC Cardiovasc Interv. 2019 Jan 14;12(1):22-32. doi: 10.1016/j.jcin.2018.10.005. PMID 30621974